CLINICAL TRIAL: NCT00326300
Title: An Open-Label, Dose-Titration, Long-Term Safety Study to Evaluate CONCERTA (Methylphenidate HCL) Extended-release Tablets at Doses of 36 mg, 54 mg, 72 mg, 90 mg, and 108 mg Per Day in Adults With Attention Deficit Hyperactivity Disorder
Brief Title: A Long-Term Safety Study to Evaluate Methylphenidate HCL Tablets at Multiple Dose Levels in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011557
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder, ADHD, Attention Deficit Disorder Adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Drug: methylphenidate hydrochloride extended-release tablets

SUMMARY:
The purpose of this study is to evaluate the long-term safety of methylphenidate HCL extended-release tablets at five dose levels in adults with Attention Deficit Hyperactivity Disorder (ADHD)

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-titration, long-term study to evaluate the long-term safety of five dose levels of methylphenidate HCL extended-release tablets, 36 mg, 54 mg, 72 mg (two 36 mg tablets), 90 mg (one 36 mg tablet plus one 54 mg tablet), and 108 mg (two 54 mg tablets) per day in adults with ADHD. At the baseline visit, all patients will initiate treatment with 36 mg of methylphenidate HCL extended-release tablets. The dose will be increased in 18 mg increments every seven days (+/-2 days) until an individualized dose is achieved. An individualized dose is achieved when there is at least a 30% improvement on the ADHD Investigator Symptoms Rating Scale (AISRS) and a Clinical Global Impression - Improvement (CGI-I) score of 1 or 2, or until the maximum dose of 108 mg is achieved. If a limiting adverse event occurs, the dose will be titrated downward by 18 mg. This dose is then the individualized dose. Once an individualized dose is achieved, patients will remain on that dose for approximately six months or one year, as assigned at the time of enrollment. Patients will be given a prescription for a one-month supply of drug and a pharmacy card at each visit. Safety assessments include monitoring adverse events, blood pressure, pulse, weight, and electrocardiograms (ECG) throughout the study. The study hypothesis is that methylphenidate HCL extended-release tablets in doses of 36 mg, 54 mg, 72 mg, 90 mg, and 108 mg per day will have an acceptable safety profile for the management of ADHD in adults.

Patients will start treatment with 36 mg extended-release tablets of methylphenidate HCL per day. The dose will be increased in 18 mg increments every 7 days (+/-2 days) until they achieve their individualized dose or reach a maximum dose of 108 mg daily. Following the patient's titration, the patient will remain on the individualized dose for approximately 6 months or one year as determined at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Investigator determined diagnosis of ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria with symptomatology from childhood to adulthood, symptoms present before age seven years and continue to meet full DSM-IV criteria at time of assessment
* Diagnosis confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) at Baseline and Adult ADHD Investigator Symptom Rating Scale (AISRS) score of 24 or greater as determined by the Investigator at Baseline
* Global Assessment of Functioning (GAF) Scale score of 41 to 60, inclusive, at Baseline
* Minimum weight of 100 lbs (45.4 kg) at Screening
* Negative urine drug test at the Screening and Baseline Visits when tested for drugs of abuse

Exclusion Criteria:

* Known to be non-responders to methylphenidate or other stimulants for the treatment of ADHD
* History of allergy, sensitivity or contraindication to methylphenidate or components of methylphenidate HCl extended-release tablets
* Coexisting medical condition or taking concomitant medication that would interfere with safe administration of methylphenidate in the Investigator's opinion
* Known structural cardiac abnormality
* Diagnosis of or family history of Tourette's syndrome, or motor or verbal tics
* History of seizures or a seizure disorder other than febrile seizures in childhood
* Glaucoma
* Uncontrolled hyperthyroidism or hypothyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2006-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Monitoring adverse events, blood pressure, pulse, and weight throughout the study; ECG at Screening, Baseline, 1 week after upward dose titration, Months 3, 6, 9, 12 or Early Termination; Laboratory tests Screening, Month 6, Month 12 or Early Termination

SECONDARY OUTCOMES:
Global Assessment of Effectiveness at titration visits, Months 3, 6, 9, 12 or Early Termination; Change from Baseline in the AISRS at titration visits, Months 3, 6, 9, 12 or Early Termination

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Derived] Adler LA, Orman C, Starr HL, Silber S, Palumbo J, Cooper K, Berwaerts J, Harrison DD. Long-term safety of OROS methylphenidate in adults with attention-deficit/hyperactivity disorder: an open-label, dose-titration, 1-year study. J Clin Psychopharmacol. 2011 Feb;31(1):108-14. doi: 10.1097/JCP.0b013e318203ea0a. PMID 21192153
- See also: Open-Label, Dose-Titration, Long-Term Safety Study of CONCERTA (36 mg, 54 mg, 72 mg, 90 mg, 108 mg) in Adults With Attention Deficit Hyperactivity Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1091&filename=CR011557_CSR.pdf